CLINICAL TRIAL: NCT03032549
Title: Short-Term Safety and Dose Effects of a Ready to Drink Pre-Workout Supplement
Brief Title: Safety of a Ready to Drink Supplement
Acronym: NB10
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas A&M University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Health Services Research
Other Study IDs: IRB2015-0754
Record Dates: First submitted 2017-01-20; First posted 2017-01-26 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2017-01

CONDITIONS: Dietary Supplements

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RTD (Experimental): 2.1 g. beta alanine, 1.3 g arginine nitrate, 200 mg caffeine, 65 mg niacin, 325 mcg folic acid, 45 mcg vitamin B12
  Interventions: Dietary Supplement: RTD
- Placebo (Placebo Comparator): dextrose and non-caloric flavoring
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: RTD — Ready to Drink Supplement
  Arms: RTD
Dietary Supplement: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This study will examine a Ready to Drink (RTD) supplement.

DETAILED DESCRIPTION:
This study will examine the short-term (7 days) characteristics of ingesting a Ready to Drink (RTD) supplement immediately prior to exercise on the blood, heart rate, blood pressure and self-reported side effects.

ELIGIBILITY:
Inclusion Criteria:

* Participants are apparently healthy and recreationally active males and females between the ages of 18 and 40

Exclusion Criteria:

* Participants are under 18 years old and above 40 years old
* Participants have a history of treatment for metabolic disease (i.e., diabetes), hypertension, hypotension, thyroid disease, arrhythmias and/or cardiovascular disease
* Participants currently use any prescription medication (birth control is allowed)
* Participants are pregnant or lactating females or plan to become pregnant within the next month
* Participants have a history of smoking
* Participants drink excessively (12 drinks per week or more)
* Participants have a recent history of creatine supplementation within 8 weeks of the start of supplementation

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2016-09-01 (Actual); Study Completion 2016-09-01 (Actual)

PRIMARY OUTCOMES:
The effects of ingesting an RTD immediately prior to exercise on the blood | 7 days
The effects of ingesting an RTD immediately prior to exercise on heart rate | 7 days
The effects of ingesting an RTD immediately prior to exercise on blood pressure | 7 days

SECONDARY OUTCOMES:
The effects of ingesting an RTD immediately prior to exercise on self-reported side effects | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Richard B Kreider, PhD, Principal Investigator — Texas A&M University

IPD SHARING:
Plan to Share IPD: No